CLINICAL TRIAL: NCT00362661
Title: Low-dose Cortisol in Chronic Posttraumatic Stress Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment: Insufficient number of patients eligible for enrollment
Sponsor: University of Zurich (Other)
Responsible Party: Dominique de Quervain, Prof. MD, University of Zurich
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PTSD-06
Record Dates: First submitted 2006-08-09; First posted 2006-08-10 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; cortisol; memory; treatment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Cortisol — Cortisol 10 mg/d for 3 months
  Other Names: Cortisol (10 mg), Galepharm, Küsnacht, Switzerland

SUMMARY:
The aim of this prospective, double-blind, placebo-controlled, cross-over study is to determine the therapeutic efficacy of low-dose cortisol for symptoms of chronic posttraumatic stress disorder.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients with chronic PTSD due to adult trauma; PTSD is diagnosed according to the DSM-IV, as measured with the CAPS
* Age between 18 and 60

Exclusion Criteria:

* History of disease states representing contraindications to glucocorticoid therapy (tuberculosis, gastritis, gastric- and duodenal ulcers, Cushing's disease, osteoporosis, hypertension, pregnancy (to exclude with a pregnancy test) and lactation, glaucoma, diabetes mellitus, thrombophilia, acute or chronic infections, hyperthyroidism, cirrhosis)
* Severe or chronic somatic diseases
* Topic glucocorticoid therapy (for large skin parts)
* Inhaled glucocorticoids
* Current psychotic, bipolar, substance-related, or severe personality disorder
* Current severe depressive disorder
* Severe cognitive impairment or a history of organic mental disorder
* Evidence of PTSD or depression immediately prior to the index trauma
* Prominent current suicidal or homicidal ideation
* Asylum seeking status
* Body weight >20% above or below normal range
* Changes in psychopharmacologic or psychotherapeutic management less than 8 weeks before start of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
CAPS CGI | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dominique de Quervain, MD, Principal Investigator — Division of Psychiatry Research, University of Zurich, Lenggstr. 31, 8032 Zurich, Switzerland; Ulrich Schnyder, MD, Principal Investigator — Department of Psychiatry, University Hospital Zurich, Culmannstrasse 8, 8091 Zürich, Switzerland
Locations (1):
- Department of Psychiatry, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Background] Aerni A, Traber R, Hock C, Roozendaal B, Schelling G, Papassotiropoulos A, Nitsch RM, Schnyder U, de Quervain DJ. Low-dose cortisol for symptoms of posttraumatic stress disorder. Am J Psychiatry. 2004 Aug;161(8):1488-90. doi: 10.1176/appi.ajp.161.8.1488. PMID 15285979